CLINICAL TRIAL: NCT05752968
Title: Elevated Levels of Antibodies to Endotoxin Core in Hemodialysis Patients With Peripheral Artery Disease
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 111064
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Endotoxemia; Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Endotoxin core antibody
MeSH Terms: conditions — Endotoxemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background

Peripheral arterial disease (PAD) and its relevant complications are more common in hemodialysis (HD) patients. The potential association regarding chronic kidney disease dysbiosis, inflammation and metabolic endotoxinemia in HD patients is unknown. A cross-sectional study will be carried out the evaluate the possible association endotoxin core antibody with asymptomatic PAD in a cohort of HD patients.

Methods

This cohort study enrolled 500 HD patients treated at a single center in Taichung city. Fasting blood samples will be collected to determine biochemical data Endotoxin core antibody levels and other related biomarkers. By the automatic oscillometric method, the ankle-brachial index (ABI) was measured. Low ABI was defined as any value < 0.9.

DETAILED DESCRIPTION:
Study Design and Patients This is a cross-sectional study involving hemodialysis patients from the hemodialysis unit of Tungs' Taichung MetroHarbor Hospital, Taiwan. A total of 500 patients over 20 years of age who receive hemodialysis with ultrapure dialysate three times weekly for at least 1 month are eligible for enrollment. We will exclude patients dialyzed with a catheter; who had an acute infection requiring hospitalization; and who had underlying malignancy or autoimmune diseases. In addition, patients who refuse to participate will be excluded. Information on participant demographics and comorbidities will be obtained from interviews and medical record reviews at the time of enrollment. Diabetes mellitus is defined by self-reported history or use of antidiabetic medications. Hypertension was defined as systolic blood pressure ≥140 mmHg, diastolic ≥90 mmHg, or use of antihypertensive agents. Pre-exisiting CVD is defined as coronary artery disease, as documented by coronary angiography or a history of myocardial infarction, class III or IV congestive heart failure, or stroke. This study will comply with the Declaration of Helsinki and will apply for approval from the Institutional Review Board of Tungs' Taichung MetroHarbor Hospital. All participants will give their written informed consent.

Laboratory Measurements Predialysis blood samples are obtained on a mid-week day. Within 30 min after sampling, the remaining blood will be centrifuged at 3,000 g for 10 min, immediately aliquoted and frozen at-70 °C until further analysis. The total serum cholesterol is measured through the reaction of cholesterol esterase/cholesterol oxidase/ peroxidase, using Hitachi 747 (Hitachi, Bohemia, NY, USA). HDL cholesterol is quantified after precipitation with polyethylene glycol at room temperature. Serum glucose concentrations are measured by the glucose oxidase method. Low-density lipoprotein cholesterol is calculated using the Friedewald formula. Total serum triglycerides are measured through the reaction of glycerol/ phosphate/oxidase and peroxidase. The serum levels of high-sensitivity C-reactive protein (hsCRP) are measured using a Behring Nephelometer II (Dade Behring, Tokyo, Japan). Serum levels of IL-6 and sCD14 are measured by a commercially available enzyme-linked immunosorbent assay (Quantikine HS Immunoassay kit, R&D System, Minneapolis, MN, USA). The LBP will be determined from serum samples and controls using standardized enzyme-linked immunosorbent assay methods (HK315-02, HyCult Biotech Inc., Uden, The Netherlands), and serum from 20 normal control subjects are used for interassay variation. Serum endotoxin core antibody will be tested using a commercially available EndoCab IgG ELISA assay (Hycult Biotech Inc., The Netherlands). In addition, serum LCN-2 (Lipocalin-2) and YKL-40 concentrations will be determined using enzyme linked immunosorbent assays

Endotoxin Measurement Endotoxin levels are measured using a Charles River Laboratories (CRL) Kinetic Chromogenic assay, Endochrome-K. A more detailed description of the methodology used has been described elsewhere [37]. Samples are thawed and diluted to 1 : 20 with a bio-dispersing agent (CRL, BD100) and heat to 75°C for 15 minutes. A standard curve (0.005 EU/mL and 5 EU/mL) is prepared using control standard endotoxin supplied by CRL. If endotoxin is detected, the samples are then reconstituted with an endotoxin-specific buffer (Charles River Endosafe BG-120) to avoid any β-glucan-related false positive reaction. A positive product control is included for each sample to eliminate the possibility of enhancement or inhibition of endotoxin measurement. The absorbance at 405 nm is measured at 30 second intervals for a total of 3600 seconds using a Biotek ELx808 plate reader. The assay reactions are held at 37°C throughout the assay period. Charles River Endosafe, EndoScan V software is used to generate a standard curve and analyze data using an onset time of 0.1 absorbance unit.

ELIGIBILITY:
Inclusion Criteria:

* A cohort of aged 20 or over, who receive hemodialysis with ultrapure dialysate three times weekly for at least 1 month.

Exclusion Criteria:

* We will exclude patients dialyzed with a catheter; who had an acute infection requiring hospitalization; and who had underlying malignancy or autoimmune diseases. In addition, patients who refuse to participate will be excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and hemodialysis (HD) for at least 1 months.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of biomarkers of endotoxin core antibody (EndoCab) levels | 1 years
  Plasma level of endotoxin core antibody (EndoCab) is a biomarkers for the risk of developing and presence of PAD

SECONDARY OUTCOMES:
Ankle Brachial Index Measurements | 1 years
  Diagnostic criterion for asymptomatic PAD
Analysis of biomarkers of IL-6 | 1 years
  The IL-6 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of sCD14 | 1 years
  The sCD14 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods assay (ELISA) methods
Analysis of biomarkers of LCN-2 (Lipocalin-2) | 1 years
  The LCN-2 (Lipocalin-2) was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of YKL-40 | 1 years
  The YKL-40 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan